CLINICAL TRIAL: NCT02610140
Title: A Randomized, Open-label, Active-controlled, Phase II Study of Intravenous Anetumab Ravtansine (BAY 94-9343) or Vinorelbine in Patients With Advanced or Metastatic Malignant Pleural Mesothelioma Overexpressing Mesothelin and Progressed on First Line Platinum/Pemetrexed-based Chemotherapy
Brief Title: Phase II Anetumab Ravtansine as 2nd Line Treatment for Malignant Pleural Mesothelioma (MPM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: ImmunoGen and MorphoSys (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15743; 2012-003650-88 (EudraCT Number)
Record Dates: First submitted 2015-11-09; First posted 2015-11-20 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — anetumab ravtansine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAY94-9343 (Experimental): Drug Anetumab ravtansine given Intravenously (IV)
  Interventions: Drug: Anetumab ravtansine (BAY94-9343)
- Vinorelbine (Active Comparator): Drug Vinorelbine given Intravenously
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Anetumab ravtansine (BAY94-9343) — Starting dose: 6.5 mg/kg administered as IV infusion over 1 h every 3 weeks until disease progression or treatment withdrawal for any reason. Dose reductions are permitted.
  Arms: BAY94-9343
Drug: Vinorelbine — Starting dose: 30mg/m^2 administered as an IV infusion over 6 to 10 min every week until disease progression or treatment withdrawal for any reason. Dose reductions are permitted per standard practise.
  Arms: Vinorelbine

SUMMARY:
The main purpose of the 15743 study is to assess efficacy and safety of anetumab ravtansine versus vinorelbine in progression free survival in patients with stage IV mesothelin overexpressing malignant pleural mesothelioma (MPM).

210 eligible patients will be randomized to receive either anetumab ravtansine every three weeks or weekly vinorelbine.

Treatment will continue until centrally confirmed disease progression or until another criterion is met for withdrawal from the study. Patients will enter follow up phase to capture safety and endpoint data as required.

Efficacy will be measured by evaluating progression free survival from randomization. Radiological tumor assessments will be performed at defined time points until the patient's disease progresses.

Blood samples will be collected for safety, pharmacokinetic and biomarker analysis. Archival or fresh biopsy tissue may also be collected for central pathology review and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of malignant pleural mesothelioma (MPM) overexpressing mesothelin
* Unresectable locally advanced or metastatic MPM after locally confirmed progression on 1st line treatment with platinum in combination with pemetrexed.
* Patients must have measurable disease
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver and renal function
* Left ventricular ejection fraction (LVEF) ≥ 50% or the lower limit of normal (LLN) according to local institution ranges of normality.

Exclusion Criteria:

* More than 1 previous systemic anti-cancer therapy line
* Patients with corneal epitheliopathy or any eye disorder that may predispose the patients to this condition at the discretion of the investigator in consultation with the ophthalmologist.
* Brain metastases, meningeal tumours or other metastases in the central nervous system
* Evidence of history of bleeding diathesis.
* Ongoing or active infection (bacterial, fungal, or viral) of National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade > 2.
* Pre-existing cardiac conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (70):
- United States (14):
  - La Jolla, California
  - Aurora, Colorado
  - Norwich, Connecticut
  - Tampa, Florida
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Bethesda, Maryland
  - Rochester, Minnesota
  - Buffalo, New York
  - New York, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Dallas, Texas
  - Houston, Texas
- Australia (5):
  - St Leonards, New South Wales
  - Woolloogabba, Queensland
  - Adelaide, South Australia
  - Richmond, Victoria
  - Nedlands, Western Australia
- Belgium (6):
  - Bruxelles - Brussel
  - Edegem
  - Ghent
  - Leuven
  - Liège
  - Sint-Niklaas
- Canada (4):
  - Calgary, Alberta
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
- Finland (3):
  - Helsinki
  - Turku
  - Vaasa
- France (6):
  - Bordeaux
  - Caen
  - Lille
  - Marseille
  - Paris
  - Pierre-Bénite
- Italy (6):
  - Pordenone, Friuli Venezia Giulia
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Monza Brianza, Lombardy
  - Turin, Piedmont
  - Siena, Tuscany
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- Poland (3):
  - Gdansk
  - Krakow
  - Szczecin
- Russia (2):
  - Omsk
  - Yekaterinburg
- Seoul, South Korea
- Spain (5):
  - A Coruña
  - Alicante
  - Barcelona
  - Madrid
  - Málaga
- Turkey (Türkiye) (6):
  - Adana
  - Ankara
  - Eskişehir
  - Istanbul
  - Malatya
  - Yenimahalle
- United Kingdom (7):
  - Plymouth, Devon
  - Maidstone, Kent
  - Leicester, Leicestershire
  - Glasgow
  - London
  - Manchester
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Kindler HL, Novello S, Bearz A, Ceresoli GL, Aerts JGJV, Spicer J, Taylor P, Nackaerts K, Greystoke A, Jennens R, Calabro L, Burgers JA, Santoro A, Cedres S, Serwatowski P, Ponce S, Van Meerbeeck JP, Nowak AK, Blumenschein G Jr, Siegel JM, Kasten L, Kochert K, Walter AO, Childs BH, Elbi C, Hassan R, Fennell DA. Anetumab ravtansine versus vinorelbine in patients with relapsed, mesothelin-positive malignant pleural mesothelioma (ARCS-M): a randomised, open-label phase 2 trial. Lancet Oncol. 2022 Apr;23(4):540-552. doi: 10.1016/S1470-2045(22)00061-4. PMID 35358455

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 315 patients were screened; of these, 67 patients were screening failures.
Groups:
- Anetumab Ravtansine (Experimental): Experimental
- Vinorelbine (Active Comparator): Active comparator
Period: Randomization and Treatment Period
Arm/Group | Anetumab Ravtansine (Experimental) | Vinorelbine (Active Comparator)
Started (Randomized) | 166 | 82
Participants Received Treatment | 163 (Safety analysis set) | 72 (Safety analysis set)
Completed | 0 | 0
Not Completed | 166 | 82
Not completed — Radiological progression | 23 | 15
Not completed — Progressive disease - radiological | 54 | 23
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Death | 7 | 1
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Adverse Event | 44 | 13
Not completed — Progressive disease - clinical | 12 | 5
Not completed — Ongoing but not completed | 9 | 2
Not completed — Not treated | 3 | 10
Period: Safety Follow-up
Arm/Group | Anetumab Ravtansine (Experimental) | Vinorelbine (Active Comparator)
Started (Safety follow-up performed) | 102 | 45
Completed | 57 | 21
Not Completed | 45 | 24
Not completed — Other | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — No follow-up | 5 | 3
Not completed — Death | 12 | 2
Not completed — Deterioration of general conditions | 15 | 5
Not completed — Withdrawal by Subject | 12 | 12
Period: Active Follow-up
Arm/Group | Anetumab Ravtansine (Experimental) | Vinorelbine (Active Comparator)
Started | 48 | 26
Completed | 0 | 0
Not Completed | 48 | 26
Not completed — Progressive disease - radiological | 30 | 22
Not completed — Death | 8 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Progressive disease - clinical | 1 | 2
Not completed — Deterioration of general conditions | 1 | 0
Not completed — Ongoing but not completed | 4 | 1
Period: Long-term Follow-up
Arm/Group | Anetumab Ravtansine (Experimental) | Vinorelbine (Active Comparator)
Started | 123 | 66
Completed | 0 | 0
Not Completed | 123 | 66
Not completed — Death | 86 | 44
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Ongoing but not completed | 30 | 17

BASELINE CHARACTERISTICS:
Population: Intent-to-treat set (ITT): all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Anetumab Ravtansine (Experimental) | Vinorelbine (Active Comparator) | Total
Number analyzed (Participants) | 166 | 82 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 37 | 103
  >=65 years | 100 | 45 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (8.1) | 65.6 (8.8) | 65.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 20 | 64
  Male | 122 | 62 | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 157 | 75 | 232
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS), [95% CI]
Description: Progression-free survival (PFS), defined as time from randomization until disease progression according to mRECIST (Modified Response Evaluation Criteria in Solid Tumors) for Malignant pleural mesothelioma (MPM) per blinded central radiology review, or death. Only descriptive analysis of OS was repeated in the follow-up period.
Time Frame: From randomization till approximately 117 PFS events observed, up to approx. 30 months (data cut-off: 31-May-2017)
Population: The primary efficacy analysis (PFS) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Anetumab Ravtansine: Test drug: 6.5 mg/kg every 3 weeks; Intravenous (IV) infusion over 1 hour
- Vinorelbine: Active comparator: 30 mg/m^2 once weekly
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
months | 4.3 [4.1 to 5.5] | 4.5 [4.1 to 5.8]
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; PFS anetumab ravtansine / vinorelbine; Test type: Superiority; p = 0.859125, Log Rank — 1-sided p-value from log-rank test (stratified by TTP on 1st line treatment). P-value is calculated based on alpha level 0.0125; Hazard Ratio (HR) = 1.215, 95% CI 2-sided [0.850 to 1,738] — Hazard ratio (anetumab ravtansine / vinorelbine) was estimated using Cox proportional hazards models with Wald CIs, stratified by Time to progression (TTP) on 1st line treatment

2. Secondary Outcome: Overall Survival (OS), [95% CI]
Description: Overall survival (OS) was defined as time from randomization until death from any cause.
Time Frame: Up to approx. 40 months (data cut-off: 06-Apr-2018) - Time from randomization until death from any cause; one-sided log-rank test stratified by time to progression (TTP) on first line treatment.
Population: The secondary efficacy analysis (OS) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
months | 9.5 [8.3 to 12.3] | 11.6 [8.6 to 13.1]
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; OS anetumab ravtansine / vinorelbine; Test type: Superiority; p = 0.655624, Log Rank — 1-sided p-value from log-rank test (stratified by TTP on 1st line treatment). Alpha spending/boundary for interim was 0.00245. Alpha boundary value for final analysis was 0.02421; Hazard Ratio (HR) = 1.072, 95% CI 2-sided [0.763 to 1.506] — Hazard ratio (anetumab ravtansine/vinorelbine) was estimated using Cox proportional hazards models with Wald CIs, stratified by TTP on 1st line treatment

3. Secondary Outcome: Objective Response Rate (ORR)
Description: A patient is a responder if the patient has a confirmed best tumor response on-study of CR (Complete response) or PR (Partial response), as determined by the central radiological reviewer per mRECIST criteria. ORR in each treatment arm was defined as the number of responders divided by the number of randomized patients. A responder was a patient who had a confirmed best tumor response on-study of CR or PR, as determined by the central radiological reviewer per mRECIST criteria.
Time Frame: up to approx. 30 months (data cut-off: 31-May-2017) - Time from randomization until death from any cause.
Population: The secondary efficacy analysis (ORR) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
percentage of participants | 8.4 [4.7 to 13.7] | 6.1 [2.0 to 13.7]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: A patient has disease control if the patient has a best tumor response on-study of CR, PR, or SD (Stable disease). DCR was defined as a percentage of patients achieving CR, PR, or SD per mRECIST criteria, as determined by the central radiological reviewer. DCR was calculated in each treatment arm as the number of patients with disease control (a best tumor response on-study of CR, PR, or SD) divided by the number of randomized patients.
Time Frame: Up to approx. 40 months (data cut-off: 06-Apr-2018) - Time from randomization until death from any cause.
Population: The secondary efficacy analysis (DCR) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
percentage of participants | 73.5 [66.1 to 80.0] | 68.3 [57.1 to 78.1]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined in responders as the time from central documentation of tumor response date of first response in the confirmation sequence) to the earlier of disease progression as determined by the central radiological reviewer, or death without centrally documented progression. A responder was a patient who had a confirmed best tumor response on-study of CR or PR, as determined by the central radiological reviewer per mRECIST criteria.
Time Frame: Up to approx. 40 months (data cut-off: 06-Apr-2018) - Time from randomization until death from any cause.
Population: The secondary efficacy analysis (DOR) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
months | 7.4 [6.0 to NA] — NA = value cannot be estimated due to censored data | 6.7 [3.0 to 10.3]

6. Secondary Outcome: Durable Response Rate (DRR)
Description: A durable responder was a responder (i.e. confirmed best tumor response on study of CR or PR) with duration of response of 180 days or more.
Time Frame: Up to approx. 40 months (data cut-off: 06-Apr-2018) - Time from randomization until death from any cause.
Population: The secondary efficacy analysis (DRR) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
percentage of participants | 7.2 [3.8 to 12.3] | 4.9 [1.3 to 12.0]

7. Secondary Outcome: Percentage of Participants With Confirmed Improvement of Symptoms Characteristic of Mesothelioma
Description: Improvement rate of symptoms characteristic of mesothelioma was defined as the number of patients with confirmed improvement of symptoms characteristic of mesothelioma (based on the MD Anderson Symptom Inventory-Malignant Pleural Mesothelioma, MDASI-MPM), divided by the number of patients evaluable for improvement of symptoms characteristic of mesothelioma.
Time Frame: up to approx. 30 months (data cut-off: 31-May-2017)
Population: The secondary efficacy analysis was performed in the ITT (Intent-to-treat) analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
percentage of participants | 22.5 [15.1 to 31.4] | 17.9 [8.9 to 30.4]
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; Anetumab ravtansine versus vinorelbine; Test type: Superiority; p = 0.244, Cochran-Mantel-Haenszel; 1-sided Cochran-Mantel-Haenszel test, stratified by TTP on 1st line treatment; Difference (%) improvement rate symptoms = 4.65, 95% CI 2-sided [-8.20 to 17.51]

8. Secondary Outcome: Time to Worsening of Symptoms Characteristic of Mesothelioma
Description: Time to worsening of symptoms characteristic of mesothelioma (TTWS) was defined in patients evaluable for assessing worsening of symptoms, as the time from randomization until the first worsening of symptoms characteristic of mesothelioma. Patients who died, were lost to follow-up, or ended (MD Anderson Symptom Inventory-Malignant Pleural Mesothelioma) MDASI-MPM assessments without confirmed worsening of symptoms were censored at the date of their last MDASI-MPM assessment with a non-missing (Composite Symptom Score) CSS.
Time Frame: up to approx. 30 months (data cut-off: 31-May-2017)
Population: The secondary efficacy analysis was performed in the ITT (Intent-to-treat) analysis set.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
days | NA [NA to NA] — value cannot be estimated due to censored data | NA [NA to NA] — value cannot be estimated due to censored data
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; Anetumab ravtansine versus vinorelbine; Test type: Superiority; p = 0.313747, Log Rank; one-sided log-rank test stratified by time to progression (TTP) on first line treatment; Hazard Ratio (HR) = 0.829, 95% CI 2-sided [0.386 to 1.779]

9. Secondary Outcome: Time to Worsening of Pain
Description: Time to worsening of pain (TTWP) was defined in patients evaluable for assessing worsening of pain, as time from randomization until the first worsening of pain. Patients who died, were lost to follow-up, or ended (MD Anderson Symptom Inventory-Malignant Pleural Mesothelioma) MDASI-MPM assessments without confirmed worsening of pain were censored at the date of their last MDASI-MPM assessment with a non-missing pain score.
Time Frame: up to approx. 30 months (data cut-off: 31-May-2017)
Population: The secondary efficacy analysis was performed in the ITT (Intent-to-treat) analysis set.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
days | 210 [127 to NA] — value cannot be estimated due to censored data | NA [85 to NA] — value cannot be estimated due to censored data
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; Anetumab ravtansine versus vinorelbine; Test type: Superiority; p = 0.378916, Log Rank; one-sided log-rank test stratified by time to progression (TTP) on first line treatment; Hazard Ratio (HR) = 0.924, 95% CI 2-sided [0.557 to 1.533]

10. Secondary Outcome: Percentage of Participants With Confirmed Improvement of Pain
Description: Improvement rate of pain was defined as the number of patients with confirmed improvement of pain (based on the "pain at its worst" item of MDASI-MPM), divided by the number of patients evaluable for improvement of pain.
Time Frame: Up to approx. 40 months (data cut-off: 06-Apr-2018) - Time from randomization until death from any cause.
Population: The secondary efficacy analysis was performed in the ITT (Intent-to-treat) analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
percentage of participants | 40.4 [30.9 to 50.5] | 32.7 [19.9 to 47.5]
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; Test type: Superiority; p = 0.214, Cochran-Mantel-Haenszel; 1-sided Cochran-Mantel-Haenszel test, stratified by TTP on 1st line treatment; Difference (%) improvement rate of pain = 6.64, 95% CI 2-sided [-9.40 to 22.68]

11. Secondary Outcome: Percentage of Participant With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as all AEs starting or worsening within the treatment period.
Time Frame: Up to approx. 55 months (data cut-off: 02-Jul-2019) - Time from randomization until 30 days after last treatment (general AEs), or further until death from any cause (selected AEs).
Population: The secondary efficacy analysis (TEAEs) was performed in the safety analysis set (SAF).
Measure: Number; unit: Percentage of participants
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 163 | 72
Percentage of participants
  Any TEAE | 99.4 | 98.6
  Any study drug-related TEAE | 88.3 | 90.3
  Treatment-emergent serious adverse events (TESAEs) | 34.4 | 34.7

12. Secondary Outcome: Number of Deaths
Description: TEAE(s) associated with a fatal outcome (CTCAE Grade 5) at the time of the data cut-off 06-Apr-2018.
Time Frame: Up to approx. 40 months (data cut-off: 06-Apr-2018) - Time from randomization until death from any cause.
Population: The secondary efficacy analysis (TEAEs) was performed in the safety analysis set (SAF).
Measure: Number; unit: Number of Deaths
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 163 | 72
Number of Deaths | 10 | 1

13. Secondary Outcome: Overall Survival (OS) - Addendum
Description: Overall survival (OS) was defined as time from randomization until death from any cause; Only descriptive analyses of OS were repeated in with the data as of the 02 JUL 2019.
Time Frame: Up to approx. 55 month (data cut-off: 02-JUL-2019) - Time from randomization until death from any cause
Population: The secondary efficacy analysis (OS) was performed in the ITT (Intent-to-treat) analysis set.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Anetumab Ravtansine | Vinorelbine
Number analyzed (Participants) | 166 | 82
months | 9.5 [8.3 to 12.3] | 11.6 [8.6 to 13.1]
Statistical Analysis 1: Comparison: Anetumab Ravtansine vs Vinorelbine; Test type: Superiority; Mean Difference (Final Values) = 9.5, 95% CI 2-sided [0.1 to 39.3]
Statistical Analysis 2: Comparison: Anetumab Ravtansine vs Vinorelbine; Test type: Superiority; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [0.0 to 35.9]

ADVERSE EVENTS:
Time Frame: Up to approx. 55 months (data cut-off: 02-Jul-2019) - Time from randomization until 30 days after last treatment (general AEs), or further until death from any cause (selected AEs).
Description: An "updated" analysis of safety:
  Treatment-emergent adverse events (TEAEs): defined as all AEs starting or worsening within the treatment period.
Groups:
- Anetumab Ravtansine (BAY94-9343): Test drug: 6.5 mg/kg every 3 weeks; Intravenous (IV) infusion over 1 hour
Arm/Group | Anetumab Ravtansine (BAY94-9343) | Vinorelbine
All-Cause Mortality (participants affected / at risk) | 126/163 | 55/72
Serious Adverse Events (participants affected / at risk) | 56/163 | 25/72
Other Adverse Events (participants affected / at risk) | 161/163 | 68/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anetumab Ravtansine (BAY94-9343) (N=163) | Vinorelbine (N=72)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (2) | 1 (2)
Pyrexia (General disorders) | 3 (3) | 3 (3)
General physical health deterioration (General disorders) | 3 (4) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (9) | 5 (6)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Scrotal mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (15) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anetumab Ravtansine (BAY94-9343) (N=163) | Vinorelbine (N=72)
Anaemia (Blood and lymphatic system disorders) | 15 (25) | 20 (42)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 5 (12)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 35 (80)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (13) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 5 (6) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 5 (5) | 0 (0)
Cataract (Eye disorders) | 9 (13) | 2 (2)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 1 (2) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 22 (26) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 3 (3) | 0 (0)
Lacrimation decreased (Eye disorders) | 6 (7) | 0 (0)
Lacrimation disorder (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Pinguecula (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 5 (6) | 0 (0)
Visual acuity reduced (Eye disorders) | 6 (7) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Corneal disorder (Eye disorders) | 65 (156) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 18 (27) | 10 (13)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (14) | 5 (5)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 29 (39) | 34 (51)
Diarrhoea (Gastrointestinal disorders) | 56 (91) | 15 (22)
Dry mouth (Gastrointestinal disorders) | 7 (8) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 13 (14) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (4) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (7) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 68 (130) | 24 (38)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 5 (6)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 34 (62) | 5 (8)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site rash (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 32 (58) | 16 (37)
Chest discomfort (General disorders) | 4 (6) | 3 (3)
Chest pain (General disorders) | 27 (31) | 13 (21)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 60 (98) | 22 (47)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 4 (4) | 0 (0)
Hyperpyrexia (General disorders) | 1 (2) | 1 (1)
Influenza like illness (General disorders) | 5 (8) | 5 (9)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 8 (13) | 5 (5)
Mass (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 3 (3)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 11 (11) | 3 (4)
Pain (General disorders) | 4 (5) | 1 (1)
Pyrexia (General disorders) | 22 (25) | 12 (14)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 3 (4) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 7 (10) | 3 (3)
Infusion site extravasation (General disorders) | 1 (1) | 1 (1)
Catheter site injury (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (5) | 3 (4)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (4) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 3 (3) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 5 (5) | 4 (4)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 5 (8)
Urinary tract infection (Infections and infestations) | 7 (9) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (5) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Oral fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (3) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 2 (2)
Tongue fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 16 (22) | 4 (4)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 20 (46) | 6 (10)
Amylase increased (Investigations) | 5 (11) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 22 (43) | 4 (4)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (5) | 2 (2)
Blood creatinine increased (Investigations) | 4 (5) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 3 (4) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 5 (5) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 11 (24) | 3 (5)
Glucose tolerance test abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (5)
Lipase increased (Investigations) | 7 (17) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (5)
Neutrophil count decreased (Investigations) | 3 (5) | 17 (41)
Platelet count decreased (Investigations) | 4 (11) | 0 (0)
Weight decreased (Investigations) | 17 (23) | 8 (12)
White blood cell count decreased (Investigations) | 2 (3) | 9 (25)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1) | 0 (0)
Hypophonesis (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 0 (0)
Waist circumference increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase decreased (Investigations) | 1 (1) | 0 (0)
Klebsiella test positive (Investigations) | 1 (1) | 0 (0)
Tear break up time decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (8) | 2 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 58 (75) | 17 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (29) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 9 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (34) | 5 (7)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (11) | 4 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (13) | 2 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (7) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 1 (1)
Asterixis (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 6 (6)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 5 (11) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 7 (9) | 1 (1)
Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 15 (17) | 5 (8)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 4 (9) | 5 (12)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 27 (52) | 5 (6)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 14 (44) | 5 (7)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (44) | 0 (0)
Polyneuropathy (Nervous system disorders) | 2 (8) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (7) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (9) | 3 (3)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (13) | 10 (10)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder trabeculation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 11 (15)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (44) | 20 (26)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermabrasion (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 9 (13) | 2 (5)
Hypotension (Vascular disorders) | 1 (2) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 6 (9)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest. Bayer will have 30-45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable). No publication of single center data should be done prior of publication if multi-center data.

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT02610140/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT02610140/SAP_001.pdf